CLINICAL TRIAL: NCT03105947
Title: Randomized Trial of Coconut Oil, Butter or Olive Oil on Blood Lipids and Metabolic Measures in Healthy Participants
Brief Title: Trial of Different Dietary Fats on Blood Lipids and Metabolic Measures in Healthy Participants
Acronym: COB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: British Broadcasting Corporation (Industry)
Responsible Party: Principal Investigator, Kay-Tee Khaw, Professor of Clinical Gerontology, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Cardiovascular Risk Factor
Keywords: lipids; dietary fats
MeSH Terms: interventions — Coconut Oil; Butter; Olive Oil

STUDY DESIGN:
Intervention Model Description: Randomized trial of different dietary fats
Who Masked: Outcomes Assessor
Masking Description: The primary outcome will be blood LDL-cholesterol, secondary outcomes, lipid profile which will be measured in a biochemistry lab by individuals who have no knowledge of the allocation to intervention arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Coconut oil (Active Comparator): 50g extra virgin coconut oil to be consumed daily for four weeks
  Interventions: Other: Coconut oil
- Butter (Active Comparator): 50g butter to be consumed daily for four weeks
  Interventions: Other: Butter
- Olive Oil (Active Comparator): 50g extra virgin olive oil to be consumed daily for four weeks
  Interventions: Other: Olive oil

INTERVENTIONS:
Other: Coconut oil — 50g extravirgin coconut oil daily for four weeks
  Arms: Coconut oil
Other: Butter — 50g butter daily for four weeks
  Arms: Butter
Other: Olive oil — 50g extra virgin olive oil daily for four weeks
  Arms: Olive Oil

SUMMARY:
This is a randomised trial in which healthy volunteers, men and women aged 50-75 years from the general community are randomized into one of three arms: participants will be provided with 50 gm extra virgin coconut oil,or 50 grams butter or 50 extra virgin olive oil to be eaten daily for a month. The key outcome is blood low density lipoprotein cholesterol concentrations and secondary outcomes blood lipid profile (total cholesterol, high density lipoprotein cholesterol, triglycerides) and anthropometric measures: weight and waist circumference. This trial is powered to detect a difference of 0.5 mmol/L LDL-cholesterol difference between the trial arms.

DETAILED DESCRIPTION:
This is a randomized trial in which healthy volunteers from the general community are randomized into one of three arms: consumption of 50 gm of extra virgin coconut oil daily OR 50gm of butter daily OR 50gm of extra virgin olive oil daily (50gm is about 2 ounces, or 2 table spoons), to be consumed over a one month period.

The research participants will be recruited from the general community through advertising (BBC).

After full informed consent, participants will attend an assessment visit and have a baseline measures of weight, height, waist circumference, blood pressure, a blood sample for assessment of blood lipids and other metabolic markers, and fill in a health questionnaire and dietary questionnaire. Participants will be randomly allocated to one of three arms: coconut oil, butter or olive oil and will be given supplies of these (portioned, or with measuring spoons) with information about daily consumption of 50 gram of one of these fats.

After one month, participants will return for follow up assessment which will include a repeat blood sample, anthropometric measures and blood pressure, and questionnaire.

Blood samples collected by venepuncture will be stored at the University of Cambridge and analysed at the Department of Clinical Biochemistry, Cambridge University Addenbrooke's Hospital.

At the end of the study, all participants will be given the individual participant results of the anthropometric measures and lipid profiles at baseline and follow up as well as the overall findings of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the trial of dietary interventions for one month within the age range

Exclusion Criteria:

* No known cardiovascular disease: heart disease or stroke; no known cancer; no known diabetes; no use of lipid lowering medication eg. statins; no contraindications to high fat diet e.g. gall bladder or other gastrointestinal condition

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
LDL-Cholesterol | after 4 weeks of the dietary fat interventions
  Blood LDL cholesterol concentrations

SECONDARY OUTCOMES:
triglycerides | after 4 weeks of the dietary fat interventions
  Blood triglycerides
HDL-Cholesterol | after 4 weeks of the dietary fat interventions
  blood HDL-Cholesterol
total cholesterol | after 4 weeks of the dietary fat interventions
  blood total Cholesterol
weight | after four weeks of the dietary fat interventions
  weight
waist circumference | after four weeks of the dietary fat interventions
  Waist circumference
Systolic Blood pressure | after four weeks of the dietary fat interventions
  systolic blood pressure

OTHER OUTCOMES:
Inflammatory markers | after four weeks of the dietary fat interventions
  Blood inflammatory markers C-Reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Kay-Tee Khaw, MBBChir, Principal Investigator — University of Cambridge
Locations (1):
- University of Cambridge, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised IPD data from the trial will be available at the end of the study with publication of the results, through contact with the principal investigator
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Once trial report published; anticipated March 2018
Access Criteria: Bona fide researchers

REFERENCES:
- [Derived] Khaw KT, Sharp SJ, Finikarides L, Afzal I, Lentjes M, Luben R, Forouhi NG. Randomised trial of coconut oil, olive oil or butter on blood lipids and other cardiovascular risk factors in healthy men and women. BMJ Open. 2018 Mar 6;8(3):e020167. doi: 10.1136/bmjopen-2017-020167. PMID 29511019